CLINICAL TRIAL: NCT07219732
Title: Boosting Exercise Adherence in Knee Osteoarthritis (BOOST-OA)
Brief Title: Boosting Exercise Adherence in Knee Osteoarthritis
Acronym: BOOST-OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD2-002-24W
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee
Keywords: exercise, physical; physical therapy, health behavior
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: In this randomized trial, 8 VHA sites will be randomized (1:1) to BOOST-OA or UC. A total of 45 participants will be enrolled at each site (n=180 per study arm). At BOOST-OA sites, behavior change initiation (concurrent) components will be delivered during the course of routine PT visits; these components are simply operationalizing "best practice" for supporting home exercise in the context of PT and not considered a new intervention. This will be followed by delivery of maintenance (sequential) components delivered virtually by a health coach; this is considered a new / experimental component of the intervention.
Who Masked: Outcomes Assessor
Masking Description: VHA sites and participants will be notified of their randomization assignment by an unblinded study team. All participant assessments will be conducted by a study team member blinded to randomization assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual PT Care (UC) (Active Comparator): UC will be delivered by trained clinicians at participating sites. The study team will provide clinicians with guidance and training to standardize core aspects of PT, aligned with best practice recommendations. Clinicians must provide enrolled Veterans with at least 4 PT visits, spaced at least weekly so that Veterans can practice home exercise and receive guidance in exercise progression. All PT visits must be completed within 3 months.
  Interventions: Behavioral: Usual PT Care (UC)
- BOOST-OA (Experimental): BOOST-OA includes components that are integrated into PT visits (concurrent), focused on behavior initiation, as well as components that occur after PT visits have ended (sequential), focused on behavior maintenance. Concurrent components will be delivered in conjunction with usual care PT visits. Clinicians must provide enrolled Veterans with at least 4 PT visits, spaced at least weekly. PT visits must be also completed within 3 months. Sequential components will be delivered by a health coach via phone or video. Health coach sessions will be conducted every other week for the first 2 months (months 4-5), monthly for an additional 3 months (months 6- 8), and every other month for the last 4 months (months 9-12; 9 total contacts). Calls will address strengthening and stretching exercises (≥3 times per week), as well as overall physical activity (e.g., minutes / steps).
  Interventions: Behavioral: BOOST-OA

INTERVENTIONS:
Behavioral: Usual PT Care (UC) — UC will be delivered by trained clinicians at participating sites. The study team will provide clinicians with guidance and training to standardize core aspects of PT, aligned with best practice recommendations. Clinicians must provide enrolled Veterans with at least 4 PT visits, spaced at least weekly so that Veterans can practice home exercise and receive guidance in exercise progression. All PT visits must be completed within 3 months.
  Arms: Usual PT Care (UC)
Behavioral: BOOST-OA — BOOST-OA includes components that are integrated into PT visits (concurrent), focused on behavior initiation, as well as components that occur after PT visits have ended (sequential), focused on behavior maintenance. Concurrent components will be delivered in conjunction with usual care PT visits. Clinicians must provide enrolled Veterans with at least 4 PT visits, spaced at least weekly. PT visits must be also completed within 3 months. Sequential components will be delivered by a health coach via phone or video. Health coach sessions will be conducted every other week for the first 2 months (months 4-5), monthly for an additional 3 months (months 6- 8), and every other month for the last 4 months (months 9-12; 9 total contacts). Calls will address strengthening and stretching exercises (≥3 times per week), as well as overall physical activity (e.g., minutes / steps).
  Arms: BOOST-OA

SUMMARY:
This project, conducted within the Department of Veterans Affairs Healthcare System (VHA), will test the effectiveness of an intervention to improve adherence to home exercise among Veterans receiving physical therapy (PT) for knee osteoarthritis (OA). The intervention, "Boosting Exercise Adherence in Knee Osteoarthritis" (BOOST-OA), has two phases. During the initiation phase (first 3 months of PT care), patients will receive tools and activities to address outcome expectations, action self-efficacy, goal-setting and monitoring. During the behavior maintenance phase (starting after PT care and continuing for 9 months), patients will receive health coaching calls that address satisfaction with outcomes, relapse prevention planning and independent monitoring. There are three main study aims: (1) examine improvements in patient outcomes, such as physical function, following BOOST-OA; (2) explore patient characteristics that lead to difference in reported improvements; and (3) interview participants and clinicians about their experience with BOOST-OA to inform future implementation.

DETAILED DESCRIPTION:
In this project, the investigators will test the effectiveness of a theoretically-informed, scalable intervention to enhance adherence to home exercise among Veterans receiving PT for knee OA. "Boosting Exercise Adherence in Knee Osteoarthritis" (BOOST-OA) includes components that address both exercise behavior initiation (conducted in conjunction with the PT episode of care) and maintenance (conducted after completion of PT care). Specifically, BOOST-OA includes: 1) Tools and activities woven into PT visits that address outcome expectations, action self-efficacy, goal-setting and monitoring (3-month behavior initiation phase) and 2) Health coaching calls that address satisfaction with outcomes, relapse prevention planning and independent monitoring (9-month behavior maintenance phase). This project is being conducted within the Department of Veterans Affairs Healthcare system (VHA). Specific aims are:

* Aim 1. Examine the effectiveness of BOOST-OA for improving physical function and other key outcomes among Veterans receiving outpatient PT for knee OA using a pragmatic cluster-randomized trial, with 8 VA PT clinics randomized to BOOST-OA vs. usual PT care (UC). Participants will be Veterans with symptomatic knee OA (n=360, 45 per site/180 per study arm). At BOOST-OA sites, behavior initiation components will be provided in conjunction with standard PT visits, and a health coach will deliver maintenance components via telehealth.
* Aim 2. Explore patient characteristics associated with differential improvement following BOOST-OA via a machine learning approach using model-based recursive partitioning. All participant characteristics, social determinants of health (SDOH), and baseline levels of study outcomes will be included in these analyses.
* Aim 3: Conduct qualitative analyses of Veteran and PT clinician experiences with BOOST-OA to inform future implementation. The investigators will conduct semi-structured interviews with Veterans (n=36 across BOOST-OA sites and a subset of UC sites) and PT clinicians delivering care to BOOST-OA participants (n=8-12) to understand acceptability, feasibility, and perceived efficacy of the program, as well as barriers and facilitators to program participation and implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of knee OA (verified from the EHR)
2. Knee pain for 3 months
3. Knee pain on most days of the previous month,
4. Average knee pain 3 (on a scale of 0-10),
5. Self-report of some difficulty with walking or stair climbing.

Exclusion Criteria:

1. Systemic rheumatic conditions, fibromyalgia, gout (knee)
2. Dementia, psychosis or active substance abuse disorder
3. Meniscus or knee ligament tear in the past 6 months
4. Lower extremity surgery in past 6 months or planned in next 9 months
5. Severe hearing or visual impairment
6. Serious / terminal illness
7. Hospitalization for a cardiovascular event, past 3 months
8. Unstable angina
9. History of ventricular tachycardia
10. Unstable chronic obstructive pulmonary disease
11. Uncontrolled hypertension (diastolic >110 mm/Hg or systolic > 200mm/Hg)
12. Stroke with moderate to severe aphasia
13. History of three or more falls in past 6 months
14. Resident of a long-term care facility
15. Other health problem that would prohibit safe participation in the study or home exercise
16. Current participation in another OA intervention study
17. Currently meeting Department of Health and Human Services physical activity recommendations
18. Completed PT for knee OA in the past year
19. Unable to speak sufficient English to participate in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale | Baseline
  The investigators selected physical function as the primary outcome because of its high importance to individuals with knee OA and its relevance for PT and exercise-based interventions. The WOMAC has been used widely in the context of clinical trials for knee OA and has well established psychometric properties including reliability, construct validity, internal consistency, and sensitivity to change in the context of behavioral interventions for knee OA. The WOMAC function subscale consists of 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale | Change from baseline to 3-months
  The investigators selected physical function as the primary outcome because of its high importance to individuals with knee OA and its relevance for PT and exercise-based interventions. The WOMAC has been used widely in the context of clinical trials for knee OA and has well established psychometric properties including reliability, construct validity, internal consistency, and sensitivity to change in the context of behavioral interventions for knee OA. The WOMAC function subscale consists of 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale | Change from baseline to 12-months (primary outcome time point)
  The investigators selected physical function as the primary outcome because of its high importance to individuals with knee OA and its relevance for PT and exercise-based interventions. The WOMAC has been used widely in the context of clinical trials for knee OA and has well established psychometric properties including reliability, construct validity, internal consistency, and sensitivity to change in the context of behavioral interventions for knee OA. The WOMAC function subscale consists of 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale | Change from baseline to 18-months
  The investigators selected physical function as the primary outcome because of its high importance to individuals with knee OA and its relevance for PT and exercise-based interventions. The WOMAC has been used widely in the context of clinical trials for knee OA and has well established psychometric properties including reliability, construct validity, internal consistency, and sensitivity to change in the context of behavioral interventions for knee OA. The WOMAC function subscale consists of 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty).
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Physical Function Subscale | Change from baseline to 24-months
  The investigators selected physical function as the primary outcome because of its high importance to individuals with knee OA and its relevance for PT and exercise-based interventions. The WOMAC has been used widely in the context of clinical trials for knee OA and has well established psychometric properties including reliability, construct validity, internal consistency, and sensitivity to change in the context of behavioral interventions for knee OA. The WOMAC function subscale consists of 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty).

SECONDARY OUTCOMES:
Patient Specific Functional Scale | Baseline
  This modified version of the Patient Specific Functional Scale will ask participants to identify one important activity they are unable to do or are having difficulty with as a result of their knee OA. They then rate their ability to perform the identified activity from 0=unable to perform to 10=able to perform at the same level as before having knee OA.
30-second Chair Stand | Baseline
  The number of times that a participant can stand up from a seated position and sit back down in 30-seconds.
2-minute Step Test | Baseline
  The number of times a participant can step in place in a 2-minute period.
WOMAC pain subscale | Baseline
  In addition to the WOMAC function subscale, the investigators will assess the WOMAC pain subscale (score range 0-20, higher scores indicate greater pain severity).
WOMAC Total Score | Baseline
  The investigators will combine WOMAC subscales to calculate a total score (score range 0-96, higher scores indicate greater pain, stiffness, and functional limitation).
Patient Specific Functional Scale | Change from baseline to 3-months
  This modified version of the Patient Specific Functional Scale will ask participants to identify one important activity they are unable to do or are having difficulty with as a result of their knee OA. They then rate their ability to perform the identified activity from 0=unable to perform to 10=able to perform at the same level as before having knee OA.
Minutes of physical activity | Baseline
  The investigators will utilize validated algorithms to calculate average minutes of light and moderate-to-vigorous physical activity per day assessed by accelerometer.
Patient Specific Functional Scale | Change from baseline to 12-months (primary outcome time point)
  This modified version of the Patient Specific Functional Scale will ask participants to identify one important activity they are unable to do or are having difficulty with as a result of their knee OA. They then rate their ability to perform the identified activity from 0=unable to perform to 10=able to perform at the same level as before having knee OA.
Patient Specific Functional Scale | Change from baseline to 18-months
  This modified version of the Patient Specific Functional Scale will ask participants to identify one important activity they are unable to do or are having difficulty with as a result of their knee OA. They then rate their ability to perform the identified activity from 0=unable to perform to 10=able to perform at the same level as before having knee OA.
Patient Specific Functional Scale | Change from baseline to 24-months
  This modified version of the Patient Specific Functional Scale will ask participants to identify one important activity they are unable to do or are having difficulty with as a result of their knee OA. They then rate their ability to perform the identified activity from 0=unable to perform to 10=able to perform at the same level as before having knee OA.
Minutes of physical activity | Change from baseline to 12-months (primary outcome time point)
  The investigators will utilize validated algorithms to calculate average minutes of light and moderate-to-vigorous physical activity per day assessed by accelerometer.
Minutes of physical activity | Change from baseline to 24-months
  The investigators will utilize validated algorithms to calculate average minutes of light and moderate-to-vigorous physical activity per day assessed by accelerometer.
30-second Chair Stand | Change from baseline to 3-months
  The number of times that a participant can stand up from a seated position and sit back down in 30-seconds.
30-second Chair Stand | Change from baseline to 12-months (primary outcome time point)
  The number of times that a participant can stand up from a seated position and sit back down in 30-seconds.
30-second Chair Stand | Change from baseline to 18-months
  The number of times that a participant can stand up from a seated position and sit back down in 30-seconds.
30-second Chair Stand | Change from baseline to 24-months
  The number of times that a participant can stand up from a seated position and sit back down in 30-seconds.
2-minute Step Test | Change from baseline to 3-months
  The number of times a participant can step in place in a 2-minute period.
2-minute Step Test | Change from baseline to 12-months (primary outcome time point)
  The number of times a participant can step in place in a 2-minute period.
2-minute Step Test | Change from baseline to 18-months
  The number of times a participant can step in place in a 2-minute period.
2-minute Step Test | Change from baseline to 24-months
  The number of times a participant can step in place in a 2-minute period.
WOMAC pain subscale | Change from baseline to 3-months
  In addition to the WOMAC function subscale, the investigators will assess the WOMAC pain subscale (score range 0-20, higher scores indicate greater pain severity).
WOMAC pain subscale | Change from baseline to 12-months (primary outcome time point)
  In addition to the WOMAC function subscale, the investigators will assess the WOMAC pain subscale (score range 0-20, higher scores indicate greater pain severity).
WOMAC pain subscale | Change from baseline to 18-months
  In addition to the WOMAC function subscale, the investigators will assess the WOMAC pain subscale (score range 0-20, higher scores indicate greater pain severity).
WOMAC pain subscale | Change from baseline to 24-months
  In addition to the WOMAC function subscale, the investigators will assess the WOMAC pain subscale (score range 0-20, higher scores indicate greater pain severity).
WOMAC Total Score | Change from baseline to 3-months
  The investigators will combine WOMAC subscales to calculate a total score (score range 0-96, higher scores indicate greater pain, stiffness, and functional limitation).
WOMAC Total Score | Change from baseline to 12-months (primary outcome time point)
  The investigators will combine WOMAC subscales to calculate a total score (score range 0-96, higher scores indicate greater pain, stiffness, and functional limitation).
WOMAC Total Score | Change from baseline to 18-months
  The investigators will combine WOMAC subscales to calculate a total score (score range 0-96, higher scores indicate greater pain, stiffness, and functional limitation).
WOMAC Total Score | Change from baseline to 24-months
  The investigators will combine WOMAC subscales to calculate a total score (score range 0-96, higher scores indicate greater pain, stiffness, and functional limitation).
Average Step Count | Baseline
  The investigators will utilize validated algorithms to calculate average steps per day assessed by accelerometer.
Average Step Count | Change from baseline to 12-months (primary outcome time point)
  The investigators will utilize validated algorithms to calculate average steps per day assessed by accelerometer.
Average Step Count | Change from baseline to 24-months
  The investigators will utilize validated algorithms to calculate average steps per day assessed by accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request, as allowable under the regulations and policies of study sponsors. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format. Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication. No data or statistical code that could lead to re-identification of individuals will be released. Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified data will be made available after study completion and as allowable by current VA policies.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.